CLINICAL TRIAL: NCT03746613
Title: Clinal Evaluation of Navigation Based Functional Ear Surgery Using Image Guided and Robotically Assisted Techniques
Acronym: EAR2OS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Vedat Topsakal (Other)
Responsible Party: Sponsor-Investigator, Prof. Vedat Topsakal, Principal Investigator, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B300201837507
Record Dates: First submitted 2018-11-12; First posted 2018-11-19 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Sensorineural Hearing Loss
Keywords: robot; Image guidance; Cochlear implantation; navigation; HEARO procedure; sensorineural hearing loss; inner ear access
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally invasive robotic cochlear implantation with HEARO (Experimental)
  Interventions: Device: HEARO

INTERVENTIONS:
Device: HEARO — Robotic system for otological procedures
  Other Names: HEARO procedure

SUMMARY:
To assess the feasibility of achieving a minimally invasive access to the inner ear through the navigation-based HEARO procedure and subsequently insert the electrode array of the cochlear implant through the access.

DETAILED DESCRIPTION:
* Demonstrate the feasibility and efficacy of performing a middle and inner ear access for cochlear implantation procedures in adults.
* Validate the procedure workflow including imaging, planning, safety assessment, image to patient registration, robotic drilling, electrode insertion and device implantation.
* Validate the system and procedure safety mechanisms.
* Collect required data for validation of safety algorithms and procedure workflow optimisation.
* Validate the HEARO system.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from profound sensorineural deafness requiring a Cochlear implant

Exclusion Criteria:

* Age under 18 years
* Pregnant women
* Anatomical anomalies of temporal bone
* Chronic otitis media with or without cholesteatoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-04-27 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
The relative ratio of successfully completed procedures where a direct access tunnel was drilled to the cochlea with the HEARO® system and the electrode was conventionally inserted through the tunnel. | Image data aquired during the procedure

SECONDARY OUTCOMES:
Number of completed middle ear access | The procedure (day 0)
Number of completed inner ear access | The procedure (day 0)
Accuracy of the drilled trajectory | Image data aquired during the procedure
Sensitivity and specificity of facial nerve monitoring | The procedure (day 0)
Measurement of the insertion angle | Image data aquired during the procedure
  Measurement of the insertion depth of the electrode into the Cochlea
Number of tip fold-overs | The procedure (day 0)
Number of Scala deviations | The procedure (day 0)
Number of complication events on (temporary) facial nerve palsy, pre and post bleeding and infection | day 0-30
Time of procedure | The procedure (day 0)
Volume of tissue removed | Image data aquired during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Antwerp, Belgium

REFERENCES:
- [Derived] Topsakal V, Heuninck E, Matulic M, Tekin AM, Mertens G, Van Rompaey V, Galeazzi P, Zoka-Assadi M, van de Heyning P. First Study in Men Evaluating a Surgical Robotic Tool Providing Autonomous Inner Ear Access for Cochlear Implantation. Front Neurol. 2022 Mar 21;13:804507. doi: 10.3389/fneur.2022.804507. eCollection 2022. PMID 35386404